CLINICAL TRIAL: NCT04754308
Title: A Study of the Incidence and Treatment of Impaired Lung Function in Patients Constituting the Target Group of Social Nurses
Brief Title: COPD and Socially Vulnerable Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Aarhus University Hospital (Other); REHPA, The Danish Knowledge Centre for Rehabilitation and Palliative Care (Other)
Responsible Party: Principal Investigator, Charlotte Suppli Ulrik, Professor, consultant, Hvidovre University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: H-20031386
Record Dates: First submitted 2021-02-10; First posted 2021-02-15 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: COPD
Keywords: Screening; Socially vulnerable patients; Social nurses
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Spirometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients referred to social nurse (Other): After obtaining informed consent, the social nurse reviews the online-questionnaire with the patient and performs a lung function examination requiring the patient to blow into a plastic tube. If a patient is identified as having obstructive reduction of lung function, they are offered a referral to a local pulmonary medicine department or GP for further investigation - regardless of whether or not they have a diagnosed or undiagnosed lung disease.
  In addition, participants are questioned about their motivation for smoking cessation and are informed of the options for this (in hospital and/or referral to the municipality).
  Interventions: Diagnostic Test: Spirometry

INTERVENTIONS:
Diagnostic Test: Spirometry — The method of examination, Spirometry, is non-invasive (i.e. not an intervention that involves penetration into the body by means of incisions or injections.). It is a routine examination and there are no risks, adverse reactions, or discomforts associated with the examination.

SUMMARY:
The trial investigates and describes the prevalence of COPD in patients who are in the social nurses' target group and investigates the effect of opportunistic screening for COPD in these vulnerable patients.

The study population is patients who have been referred to a social nurse at hospitals in the Capital Region, Central Denmark Region and Region Zealand of Denmark during the inclusion period, and monitor them for up to 5 years in order to investigate variables that are significant in terms of the patients' treatment, hospitalisations, and mortality in relation to COPD.

Our hypothesis is that there will be a higher incidence of COPD among those patients with whom the social nurses have contact than in the general population.

DETAILED DESCRIPTION:
The study consists of two sub-studies: A a descriptive cross-sectional study "The prevalence of COPD in patients who are in the social nurses' target group" followed by study B a cohort study "The effect of opportunistic screening for COPD in patients who are in the social nurses' target group", based on a closed cohort.

People in the lower social classes are at increased risk of developing COPD due to their lifelong accumulation of risk factors, such as smoking, passive smoking and the influence of lifestyle and the environment.

In the group with the socially vulnerable individuals, 70% are smokers compared to 18% in the general Danish population. The socially vulnerable individuals are defined here as people affected by homelessness, drug abuse, harmful alcohol consumption, mental illness and poverty. Despite the socially vulnerable group having an over-consumption of general practice visits, 25% of the patients in the social nurses' target group state that they do not have contact with or use their own doctor.

Our hypothesis is therefore that there will be a higher incidence of COPD among those patients with whom the social nurses have contact than in the general population.

Purpose: To investigate and describe the prevalence of COPD in patients who are in the social nurses' target group and to investigate the effect of opportunistic screening for COPD in these vulnerable citizens.

Data collection:

Baseline data from the cross-sectional study are derived from lung function measurement and REDCap online-questionnaires completed on inclusion.

The data from the cohort study regarding disease burden and hospital visits originates from the national patient registry (LPR) and mortality data is retrieved from the Danish Register of Causes of Death. Data regarding redeemed prescriptions for COPD medicine originates from the Prescription Database. The patients' connection to the job market and income status are based on extracts from RAS (Registry-based Labour Force Statistics), which is administered by Statistics Denmark. Data regarding the highest acquired education (HFAUDD) is from Statistics Denmark.

Variables:

There will be collected the following variables at inclusion: information on demographics, lung function, selv-reported information on: risk factors, socioeconomic variables and symptoms of lung disease. Moreover register data on socioeconomic status, morbidity, physical health by Charlson score, mortality, hospital visits and prescriptions for COPD Medicine will be retrieved after 5 years follow-up.

Sample size:

To detect a difference between the patient group and the Danish population of minimum 100% a total of 511 participants are needed in the study (power of 80%, p-values=0,05, an estimated COPD prevalence of 4,3% in the Danish population).

The collected data will be kept in accordance to the Data Protection Agency guidelines. The studies are carried out in accordance with the principles of the Helsinki Declaration.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Able to speak and understand Danish to such an extent that informed consent can be obtained

Exclusion Criteria:

* Not having a Danish civil registration number, since foreign patients do not have free access to examinations and medical treatment, and cannot be followed up in the national patient registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 513 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2024-04-18 (Actual); Study Completion 2024-04-18 (Actual)

PRIMARY OUTCOMES:
Prevalence of obstructive lung function reduction in patients in the social nurses' target group | Baseline
Distribution of diagnosed and undiagnoses COPD in patients | Baseline
Numbers of patients diagnosed with obstructive lung function that are subsequently examined at a pulmonary medicine outpatient clinic/GP | Baseline
Prevalence of patients diagnosed with COPD after screening | Baseline
Does opportunistic screening by social nurses impact on the number of hospital visits? | Follow-up 5 years from inclusion
  The outcome is number of outpatient and acute visits with a-diagnosis related to COPD for 3 groups of patients: The group with undiagnosed COPD at inclusion who were investigated, and the group with undiagnosed COPD at inclusion who did not want investigation compared with the group of patients with already diagnosed COPD at inclusion (control group).
Does opportunistic screening by social nurses affect medication consumption in connection with the treatment of COPD? | Follow-up 5 years from inclusion
  The outcome is redeemed prescriptions for COPD medication among the 2 groups of patients: The group with undiagnosed COPD at inclusion compared with the group of patients with already diagnosed COPD at inclusion (control group).

SECONDARY OUTCOMES:
Prevalence of patients who smoke and wish to stop smoking | Baseline
Prevalence of patients with impaired lung function who have a desire to stop smoking | Baseline
Prevalence of patients who want to quit smoking and accept the smoking cessation offers. | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Nina Brünés, Study Chair — Amager and Hvidovre Hospital, Patientforloeb; Charlotte Ulrik, Principal Investigator — Amager and Hvidovre Hospital, Medical Department
Locations (10):
- Denmark (10):
  - Århus Universitetshospital, Aarhus
  - Bispebjerg and Frederiksberg Hospital, Copenhagen
  - Copenhagen University Hospital Rigshospitalet, Copenhagen
  - Herlev and Gentofte Hospital, Copenhagen
  - Regionshospitalet Horsens, Horsens
  - Hvidovre Hospital, Hvidovre
  - Sjællands Universitetshospital Køge og Roskilde, Køge
  - Nykøbing Falster Sygehus, Nykøbing Falster
  - Bornholm Hospital, Rønne
  - Næstved-Slagelse-Ringsted Hospital, Slagelse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brunes N, Lindstroem MB, Ulrik CS, Andersen O, Lisby M, Godtfredsen NS, Hansen TL, Pisinger C, Graven V, Marsaa K, Thomsen LH. Opportunistic screening for COPD among socially marginalized patients. BMC Pulm Med. 2024 Mar 5;24(1):113. doi: 10.1186/s12890-024-02927-9. PMID 38443835